CLINICAL TRIAL: NCT03298139
Title: THE INFLUENCE OF GRAVITY ON TARGET CUEING DURING VISUAL SEARCH USING AUGMENTED REALITY
Brief Title: THE INFLUENCE OF GRAVITY
Acronym: ARGuide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Basic Science
Other Study IDs: 16-115
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- parabolic flights (Experimental): parabolic flights in normogravity (1g), hypergravity (1.8g) and microgravity (0g).
  Interventions: Other: 3 levels of gravity (1G, 1.8G, 0G).

INTERVENTIONS:
Other: 3 levels of gravity (1G, 1.8G, 0G). — healthy volunteers will experience 3 levels of gravity (1G, 1.8G, 0G).

SUMMARY:
Although most ground studies showed that an egocentric reference frame better supports spatial orientation, it is not proven it will be the same during weightlessness.

Although it might justify that visuomotor performance will be better supported by egocentric target cueing under altered gravity conditions, the fact that exocentric target cueing induces less head movements and called for least attentional and physiological workload could be the key factors for a more efficient task localization process. Moreover, weightlessness can induce spatial disorientation, which can be additionally influenced by the intrinsic and extrinsic spatial reference frames (Gurfinkel et al., 1993; Glasauer & Mittelstädt, 1997, 1998; Harm et al., 1998; Lipshits et al. 2005). We expect that during weightlessness the workload will be the key factor and thus we hypothesize that an exocentric target cueing will outperform egocentric target cueing.

To test this hypothesis, and find out which presentation scheme for target cueing (EGO, EXO, ED) contributes most to an efficient visual search, performance to a visuomotor task will be evaluated during parabolic flights in normogravity (1g), hypergravity (1.8g) and microgravity (0g). The visuomotor performance will be assessed by a multi-directional tapping task as defined by ISO9241-9, which requests for motor responses by aimed pointing movements. Besides analyzing the pointing performance, different workload indices will be additionally assessed to evaluate the effort spent on visuomotor coordination. The attentional workload will be evaluated by the performance of a secondary task (visual reaction-time task), which needs to be conducted in parallel to the visuomotor task. Furthermore, the workload will be also assessed subjectively by the NASA TLX rating scale and physiologically, by analyzing the heart rate variability (HRV).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 67
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Pregnant women

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
visuomotor performance | baseline
  The visuomotor performance will be assessed by a multi-directional tapping task as defined by ISO9241-9, which requests for motor responses by aimed pointing movements.
common external display guidance method (ED) | baseline
  common external display guidance method (ED) and exocentric "in-view" cueing (EXO), using common guidance method with an external display (ED) as a control condition

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No